CLINICAL TRIAL: NCT03713242
Title: A Single-center, Open-label, Single-dose, Phase 1 Study to Evaluate the Pharmacokinetics of ACT-541468 in Subjects With Mild, Moderate, and Severe Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics of ACT-541468 in Subjects With Mild, Moderate, and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-078-112; NCT03686995 (obsolete NCT alias)
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: prospective, single-center, open-label, single-dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: ACT-541468 in subjects with mild hepatic impairment (Experimental): Single oral dose administered on Day 1.
  Interventions: Drug: ACT-541468 25 mg
- Group B: ACT-541468 in subj. with moderate hepatic impairment (Experimental): Single oral dose administered on Day 1.
  Interventions: Drug: ACT-541468 25 mg (or 10 mg depending on interim results)
- Group C: ACT-541468 in subjects with severe hepatic impairment (Experimental): Single oral dose administered on Day 1.
  Interventions: Drug: ACT-541468 25 mg (or 10 mg depending on interim results)
- Group D: ACT-541468 in healthy subjects. (Experimental): Single oral dose administered on Day 1.
  Interventions: Drug: ACT-541468 25 mg (or 10 mg depending on interim results)

INTERVENTIONS:
Drug: ACT-541468 25 mg — Administered as a tablet.
  Arms: Group A: ACT-541468 in subjects with mild hepatic impairment
Drug: ACT-541468 25 mg (or 10 mg depending on interim results) — Administered as a tablet.
  Arms: Group B: ACT-541468 in subj. with moderate hepatic impairment; Group C: ACT-541468 in subjects with severe hepatic impairment; Group D: ACT-541468 in healthy subjects.

SUMMARY:
This is a prospective, single-center, open-label, single-dose, Phase 1 study, to assess the effect of mild, moderate, and severe hepatic impairment due to liver cirrhosis on the pharmacokinetics of ACT-541468.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male and female subjects aged between 18 and 75 years (inclusive) at screening.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use (from screening, during the entire study, and for at least one month after last study treatment intake) a highly effective method of contraception, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential.
* Body mass index of 18.0 to 35.0 kg/m2 (inclusive) at screening.
* For healthy subjects: Normal renal function confirmed by a creatinine clearance at screening according to Cockroft and Gault adjusted to age of:

  1. ≥ 80 mL/min/1.73 m2 for subjects ≤ 50 years of age.
  2. ≥ 70 mL/min/1.73 m2 for subjects 51-60 years of age.
  3. ≥ 60 mL/min/1.73 m2 for subjects 61-75 years of age.
* For subjects with hepatic impairment: Degree of liver function impairment due to liver cirrhosis according to the Child-Pugh classification:

  1. Group A: Mild hepatic impairment, Child-Pugh score 5-6.
  2. Group B: Moderate hepatic impairment, Child-Pugh score 7-9.
  3. Group C: Severe hepatic impairment, Child-Pugh score 10-15.

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* For subjects with hepatic impairment: History of major medical or surgical disorders, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment except for those related to liver cirrhosis (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* For healthy subjects:

  1. History of alcoholism or drug abuse within the 3-year period prior to screening.
  2. Relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (AEs) | From study treatment administration up to EOS (duration: up to 4 days)
Treatment-emergent serious adverse events (SAEs) | From study treatment administration up to EOS (duration: up to 4 days)

OTHER OUTCOMES:
Plasma pharmacokinetics: AUC(0-t) | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: AUC(0-inf) | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: AUC(0-24) | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: Cmax | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: Tmax | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: T1/2 | At various timepoints (duration: up to 4 days)
Plasma pharmacokinetics: Cu/C (extent of plasma protein binding) | At various timepoints (duration: up to 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger B, Dingemanse J, Sabattini G, Delahaye S, Duthaler U, Muehlan C, Krahenbuhl S. Effect of Liver Cirrhosis on the Pharmacokinetics, Metabolism, and Tolerability of Daridorexant, A Novel Dual Orexin Receptor Antagonist. Clin Pharmacokinet. 2021 Oct;60(10):1349-1360. doi: 10.1007/s40262-021-01028-8. Epub 2021 May 18. PMID 34002356